CLINICAL TRIAL: NCT04626570
Title: Impact of a Phone-based Cognitive and Behavioral Therapy on Food Addiction in Patients With Severe or Morbid Obesity
Acronym: ADALOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR190068; 2019-A02773-54 (Other: IdRCB)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Food Addiction
Keywords: obesity; food addiction; binge eating disorder; psychiatric disorders; addictive disorders; obesity-specific quality of life; metabolic syndrome; diabetes; dyslipidemia; hypertension; hepatic cytolysis; cognitive and behavioral therapy
MeSH Terms: conditions — Obesity; Food Addiction; Binge-Eating Disorder; Mental Disorders; Metabolic Syndrome; Diabetes Mellitus; Dyslipidemias; Hypertension | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive and Behavioural Therapy plus Management as usual (Experimental): 12 sessions of CBT during 18 weeks AND management of obesity with nutritional and dietary treatment as usual
  Interventions: Other: Cognitive and Behavioral Therapy
- Management as usual (No Intervention): management of obesity with nutritional and dietary treatment as usual

INTERVENTIONS:
Other: Cognitive and Behavioral Therapy — 12 sessions of CBT using a standardized approach
  Arms: Cognitive and Behavioural Therapy plus Management as usual

SUMMARY:
Morbid or severe obesity is a chronic pathology of multifactorial etiology that affects 4.3% of the French population. In these patients, eating disorders are frequent and must be managed as they are considered risk factors with poorer weight prognosis and lower quality of life.

Some authors have proposed that the concept of food addiction (i.e., the existence of an addiction to certain foods rich in sugar, fat and/or salt) may make it possible to identify, among obese patients, a subgroup of patients that is more homogeneous in terms of diagnosis and prognosis.

Food addiction is common in obese patients and is associated with higher levels of depression, anxiety, impulsivity, emotional eating and poorer quality of life. Nevertheless, we do not know the impact of managing this addiction on the future of these patients (food addiction, weight, comorbidities, quality of life). Telephone-based cognitive behavioral therapy intervention (Tele-CBT) is a treatment of choice for addictions, but there are inequalities in access to this treatment (distance between home and hospital, limited local resources of caregivers, constraints in patient availability) which require the therapeutic framework to be adapted to these constraints. A short Tele-CBT program has demonstrated its effectiveness in reducing bulimic hyperphagia in these patients (Cassin et al. 2016), but its effectiveness on food addiction, Body Mass Index and the evolution of metabolic complications related to obesity is still unknown. The evaluation of this program was limited to 6 weeks (American study), and we do not know if these results can also be extrapolated to France.

The main hypothesis of this study is that in patients suffering from severe or morbid obesity and with food addiction, the performance of tele-CBT (intervention group: 12 sessions for 18 weeks) will be accompanied by a significant medium-term decrease in the prevalence of food addiction compared to usual management (control group).

DETAILED DESCRIPTION:
Morbid or severe obesity is a chronic pathology of multifactorial etiology that affects 4.3% of the French population. In these patients, eating disorders are frequent and must be managed as they are considered risk factors with poorer weight prognosis and lower quality of life.

Some authors have proposed that the concept of food addiction (i.e., the existence of an addiction to certain foods rich in sugar, fat and/or salt) may make it possible to identify, among obese patients, a subgroup of patients that is more homogeneous in terms of diagnosis and prognosis.

Food addiction is common in obese patients and is associated with higher levels of depression, anxiety, impulsivity, emotional eating and poorer quality of life. Nevertheless, we do not know the impact of managing this addiction on the future of these patients (food addiction, weight, comorbidities, quality of life). Telephone-based cognitive behavioral therapy intervention (Tele-CBT) is a treatment of choice for addictions, but there are inequalities in access to this treatment (distance between home and hospital, limited local resources of caregivers, constraints in patient availability) which require the therapeutic framework to be adapted to these constraints. A short Tele-CBT program has demonstrated its effectiveness in reducing bulimic hyperphagia in these patients (Cassin et al. 2016), but its effectiveness on food addiction, Body Mass Index and the evolution of metabolic complications related to obesity is still unknown. The evaluation of this program was limited to 6 weeks (American study), and we do not know if these results can also be extrapolated to France.

The main hypothesis of this study is that in patients suffering from severe or morbid obesity and with food addiction, the performance of tele-CBT (intervention group: 12 sessions for 18 weeks) will be accompanied by a significant medium-term decrease in the prevalence of food addiction compared to usual management (control group).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI ≥35kg/m² (morbid or severe obesity)
* First appointment to a physician specialized in nutrition
* "Food addiction diagnosis" according to the YFAS 2.0
* Affiliated to the French national health service
* Consent signed

Exclusion Criteria:

* Difficulties in understanding the self-administered questionnaires, including illiteracy
* Impossibility to participate to the CBT sessions (i.e., no phone, scheduled unavailability)
* Not eligible for CBT (i.e., cognitive disorders, hearing disorders)
* Antecedent of monogenic or oligogenic obesity (MC4R mutation)
* Severe alcohol use disorder (at least 6 out of 11 DSM-5 criteria for alcohol use disorder)
* Current medication with a significant adverse effect on eating behavior (i.e., lithium, neuroleptic/antipsychotic)
* Discrepancy between self-administered questionnaires and the clinical interview conducted prior to inclusion (for the assessment of food addiction diagnosis).
* Condition associated with important weight variations (i.e., oedema related to severe cardiac insufficiency, renal insufficiency, hepatic insufficiency with cirrhosis, exudative enteropathy)
* Participation to another psychological or pharmacological interventional study that could impact our primary or secondary outcomes
* Wearing a pace-maker or metal prosthesis
* Person under tutorship or curatorship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Percentage of patients without food addiction | 18 weeks after randomization
  Yale Food Addiction Scale 2.0 (food addiction is defined by the existence of at least 2 out of 11 criteria for food addiction and associated emotional distress)

SECONDARY OUTCOMES:
Evolution of Percentage of patients without food addiction during follow-up | From baseline, up to 9 months
  Yale Food Addiction Scale 2.0 (food addiction is defined by the existence of at least 2 out of 11 criteria for food addiction and associated emotional distress)
Evolution of number of criteria for food addiction | From baseline, up to 9 months
  Yale Food Addiction Scale 2.0 (food addiction is defined by the existence of at least 2 out of 11 criteria for food addiction and associated emotional distress)
Weight/BMI evolution | From baseline, up to 9 months
  Weight and height measurement
Evolution of the waist-to-hip ratio | From baseline, up to 9 months
  Waist and hip measurement
Evolution of Body Composition | From baseline, up to 9 months
  Impedancemetry
Existence and evolution psychiatric and addictive disorders | From baseline, up to 18 weeks
  Mini International Neuropsychiatric Interview 5.0.0 (MINI 5.0.0)
Existence and evolution of depression | From baseline, up to 9 months
  Beck Depression Inventory (BDI)
Existence and evolution of bulimic hyperphagia | From baseline, up to 9 months
  Binge Eating Scale (BES)
Existence and evolution of an alcohol use disorder | From baseline, up to 9 months
  Alcohol Use Disorder Inventory Test (AUDIT)
Existence and evolution of a Smoking Disorder | From baseline, up to 9 months
  Fagerström Test for Nicotine Dependence (FTND)
Existence and evolution of food cravings | From baseline, up to 9 months
  Food Cravings Questionnaire-Trait-reduced (FCQ-T-r)
Existence and evolution of emotional eating | From baseline, up to 9 months
  Dutch Eating Behavior Questionnaire (DEBQ)
Evolution of quality of life | From baseline, up to 9 months
  Quality of Life, Obesity and Dietetics (QOLOD)

CONTACTS AND LOCATIONS:
Overall Officials: Paul BRUNAULT, MD, Study Director — University Hospital, Tours
Locations (9):
- France (9):
  - Department of endocrinology-diabetology-nutrition, University Hospital, Angers, Angers
  - Nutrition Department, University Hospital, Brest, Brest
  - Transversal Clinical Nutrition Unit, University Hospital, Caen, Caen
  - Transversal Nutrition Unit, Hospital, Cherbourg, Cherbourg
  - Nutrition Department, University Hospital, Nantes, Nantes
  - Department of Internal Medicine, Endocrinology and Metabolic Diseases, University Hospital, Poitiers, Poitiers
  - Endocrinology, diabetology and nutrition department, University Hospital, Reims, Reims
  - Endocrinology, diabetology and nutrition department, University Hospital, Rennes, Rennes
  - Metabolic and nutritional exploration, University Hospital, Tours, Tours